CLINICAL TRIAL: NCT01925339
Title: Esthetic Outcomes of Immediately Placed Implants Receiving Immediate Provisionalization and Delayed Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Collegiate Professor of Periodontics and Professor of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00070747
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Tooth Diseases; Tooth Extraction; Dental Implant
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test (immediate restoration) (Experimental): Test (immediate restoration): immediate restoration will be placed on immediately placed implants.
  Interventions: Device: Test (immediate restoration)
- Control: delayed restoration (Experimental): Control: delayed restoration: immediate placed implants will be restored at 4 months.
  Interventions: Device: Control: delayed restoration

INTERVENTIONS:
Device: Test (immediate restoration) — Test (immediate restoration)
  Arms: Test (immediate restoration)
Device: Control: delayed restoration — Control: delayed restoration
  Arms: Control: delayed restoration

SUMMARY:
The purpose of this study is to compare two different timings of restoring dental implants that are placed right after tooth extraction: The test group will have the provisional crown placed at the time of implant placement. The control group will have the tooth removed and the implant placed at the same appointment but restorations placed after 4 months. Both procedures currently are accepted methods for replacing missing teeth but direct comparisons of the two procedures are lacking. The results of this study should aid clinicians in selecting the best timing for restoring implants for their patients. The hypothesis is that immediate restoration might increase aesthetic outcomes, e.g. less mucosal recession.

DETAILED DESCRIPTION:
A single center, randomized controlled, parallel-arm study is planned to investigate esthetic outcomes after immediate placement and restoration in the esthetic zone. Forty adult patients who have a hopeless maxillary anterior or premolar tooth, with intact adjacent teeth will be enrolled. A signed written informed consent will be obtained after he or she has been given verbal and written information describing the nature and duration of the study. Subjects will not be screened or treated until an informed consent has been obtained. Patient information will be protected according to the privacy regulations of the Federal Health Insurance Portability and Accountability Act of 1996 (HIPAA).

The enrolled patients will be randomly placed into one of two treatment groups, immediate implant placement (IIP) and restoration group (IR) or the IIP + delayed restoration group (DR). For all patients, the hopeless tooth will be extracted atraumatically and an implant placed immediately. The decision will be made randomly to either restoring the implant immediately (Test group) with a provisional crown or restoring the implant at 4 months after implant placement (Control group). Outcome analyses will be performed until approximately 1-year after the implant surgery and primarily evaluate clinical and radiographic parameters to determine the esthetic outcomes of immediately restored IIP implants, in comparison to those immediately placed but restored in a delayed approach.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 21 or older
* A minimum dentition of 20 permanent teeth (including natural rooted teeth or dental implants; pontic of a fixed bridge is not considered a tooth)
* A maxillary premolar, canine, lateral incisor or central incisor with a hopeless prognosis
* Presence of adjacent teeth and enough clearance for an implant crown
* Presence of sufficient bone apical to the root apex of the hopeless tooth

Exclusion Criteria:

Systemic criteria:

* Current heavy smokers (>10 cigarettes per day) or heavy smokers who quitted less than 1 year
* Pregnant or plan to get pregnant or lactating mothers
* Diseases of the immune system or any medical condition that may influence the outcome (uncontrolled diabetes (HbA1c >7), neurologic or psychiatric disorders, systemic infections, …)
* Radiation therapy in the head and neck area within 3 years
* Current use of oral bisphosphonates for >3 years
* History of IV bisphosphonates use
* Other medical conditions that may contradict an implant surgery

Intraoral criteria:

* Area of study is adjacent to an existing implant
* Acute infection at/or adjacent to the extraction site (e.g., sinus tract, swelling, etc.)
* Observable gingival changes due to use of medications such as calcium antagonists, anticonvulsives, immunosuppressives, anti-inflammatory medications, etc.)
* Untreated deep carious lesions or defective restorations that can potentially exacerbate during the course of the experiment
* Uncontrolled periodontal disease
* Poor oral hygiene (>20% FMPS)

CBCT criteria:

• More than 4 mm of buccal plate dehiscence is present on CBCT scans

Intraoperative criteria:

• More than 4 mm of buccal plate dehiscence is present once the tooth is extracted

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS, MSD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test (Immediate Restoration) | Control: Delayed Restoration
Started | 20 | 20
Completed | 18 | 20
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Immediate Restoration) | Control: Delayed Restoration | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (12.4) | 57.9 (15.0) | 59.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 20 | 20 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 20 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Mucosal Recession Change
Description: Mucosal level change from baseline to one year was primarily determined by an imaginary line connecting the gingival margin of the adjacent teeth. This was measured in millimeters.
Time Frame: Baseline, 1 year
Population: Two subjects withdrew from the study prior to the 1 year time point. Therefore, no data was analyzed for these two subjects.
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Test (Immediate Restoration) | Control: Delayed Restoration
Number analyzed (Participants) | 18 | 20
milimeters | 0.1 (0.9) | 0.1 (0.7)

2. Secondary Outcome: Radiographic Marginal Bone Level Change
Description: Mean of mesial and distal marginal bone level changes measured by standard radiographs using customized device. This was measured in millimeters.
Time Frame: Baseline, 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Test (Immediate Restoration) | Control: Delayed Restoration
Number analyzed (Participants) | 18 | 20
milimeters | 0.8 (0.7) | 0.8 (0.6)

ADVERSE EVENTS:
Time Frame: Fifteen months for each subject.
Arm/Group | Test (Immediate Restoration) | Control: Delayed Restoration
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 13/20 | 12/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (Immediate Restoration) (N=20) | Control: Delayed Restoration (N=20)
Issues related to tooth #30 (General disorders) | 0 (0) | 1 (1) — One subject had the crown on tooth #30 come off.
Appendix removed (Surgical and medical procedures) | 1 (1) | 0 (0) — One subject had his appendix surgically removed.
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — One subject was treated for atrial fibrillation.
Asthma attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — One subject reported being treated by her primary care physician for asthma-related symptoms.
Bad taste in mouth (General disorders) | 0 (0) | 2 (2) — Two subjects reported having a bad taste in her mouth.
Bone grafting material at implant site (General disorders) | 0 (0) | 1 (1) — One subject had extra bone grafting particles at implant site.
Dental cavity (General disorders) | 1 (1) | 1 (1) — Two subjects reported having to have dental cavity fixed.
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — One subject reported going to a doctor to be tested for a blood disorder.
Falls (General disorders) | 0 (0) | 2 (2) — Two subjects reported accidentally falling and having to see their primary care physicians.
Deep vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — One subject reported being treated for a deep vein thrombosis.
Dehydration (General disorders) | 1 (1) | 0 (0) — One subject reported being treated for dehydration.
Gastrointestinal problems (Gastrointestinal disorders) | 1 (1) | 1 (1) — One subject reported being treated for diarrhea. One subject reported being treated for diverticulitis.
Tooth sensitivity (General disorders) | 1 (1) | 1 (1) — Two subjects reported having dental sensitivity around non-study teeth.
Tooth abscess (General disorders) | 1 (1) | 0 (0) — One subject had a tooth abscess on a non-study tooth.
Exudate at implant site (General disorders) | 3 (3) | 3 (3) — Exudate (pus) was noted at implant site.
Gum tissue tenderness (General disorders) | 2 (2) | 0 (0) — Two subjects reported having gum tissue tenderness.
Ingrown toe nail (Surgical and medical procedures) | 0 (0) | 1 (1) — One subject had an ingrown toe nail surgically removed.
Healing abutment (General disorders) | 3 (3) | 2 (2) — Healing abutment screw became loose.
Exposed implant (General disorders) | 1 (1) | 0 (0) — One subject's implant perforated the buccal plate.
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0) — One subject was treated for a kidney stone.
Poison ivy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — One subject reported being treated for poison ivy.
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) — One subject reported having multiple flu-like symptoms.
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One subject reported seeing her primary care physician for sports-related shoulder pain.
Shingles (Immune system disorders) | 1 (1) | 0 (0) — One subject reported being treated for shingles.
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — One subject reported being treated for a sinus infection.
Gum tissue inflammation (General disorders) | 1 (1) | 0 (0) — One subject had a lot of gum tissue inflammation at the site of the implant.
Swelling (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — One subject reported being treated for swelling in her hands and feet.
Issues with temporary crown (General disorders) | 2 (3) | 0 (0) — Two subjects had minor issues with their temporary crowns.
Tissue impingement (General disorders) | 0 (0) | 1 (1) — One subject's healing abutment was impinging on the adjacent tissue.
Broken tooth (General disorders) | 0 (0) | 1 (1) — One subject reported having a broken non-study tooth.
Tissue trauma (General disorders) | 0 (0) | 1 (1) — One subject had tissue trauma from eating at the site of the implant.
Twisted ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Two subjects reported twisting their ankles and needing to be seen by their physicians.
Urinary track infection (Renal and urinary disorders) | 1 (1) | 1 (1) — Two subjects reported being treated for urinary track infections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT01925339/Prot_SAP_000.pdf